CLINICAL TRIAL: NCT03994952
Title: Comparison of a Non-linear Analysis of Balance During the mBESS to the Sway Balance Application
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0454-19-EP
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: Balance, postural; Non-linear dynamics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Uninjured Physically Active Young Adults: This is a group of physically active, and currently uninjured young adults. They will complete a single balance assessment, the modified balance error scoring system protocol, as outlined by the Sway Balance application.
  There is no comparison group for this investigation.
  Interventions: Device: Sway Balance Application; Device: Balance Tracking Systems

INTERVENTIONS:
Device: Sway Balance Application — Participants complete the modified Balance Error Scoring System as prompted on and iPad mini. It has 5 balance stances, double limb stance, right tandem, left tandem, right single, and left single leg balance for 20 seconds each. This will only be used as measurement, not an intervention.
Device: Balance Tracking Systems — This is a force platform. Center of pressure data will be measured and recorded while participants are completing the modified Balance Error Scoring System. This will only be used as measurement, not an intervention.

SUMMARY:
In order to determine equivalency of the Avert Sample Entropy algorithm's ability to be sensitive to different balance conditions, participants will complete the modified balance error scoring system (mBESS) while standing on a portable force platform. Human-rated errors during the mBESS conditions will be recorded, in addition to measuring balance using the Sway app. These will be compared for levels of agreement and direction of bias using Bland-Altman analyses.

DETAILED DESCRIPTION:
This investigation will utilize a single session of data collection, which should last no longer than 10 minutes per participant. During this session, the investigators will obtain informed consent, and then the participant will complete a balance test comprised of five, 20-second trials.

The testing procedures are as follows. All participants will perform the mBESS protocol as outlined by the Sway Balance Application. This protocol consists of a total of 5 balance trials, each being 20 seconds in duration. Every balance trial is completed with the eyes closed. Each trial has a different stance configuration: eyes closed feet together, eyes closed right tandem stance (one foot in front of the other, touching the toe to the heel), eyes closed left tandem stance, eyes closed right foot balance, eyes closed left foot balance.

During the test, the participant will hold an iPad mini to their torso, right in front of their sternum and follow the audio prompts to begin balancing and when the balance trial is over. The participant will be given instructions that they can change their stance if they lose their balance, and take a compensatory step if they need it to catch their balance. The participant will be standing on a Balance Tracking Systems force platform for each test, in order to capture an additional objective measurement of their balance. The participant will be asked to ensure they have at least one foot in contact with the plate during each trial.

If a participant should step off of the force platform during an individual trial, the participant will re-do that balance condition to ensure that each participant has one complete 20-second trial that has a score from the Sway app, as well as a full 20-second dataset from the force platform.

The PI will also perform BESS scoring during each trial, and count errors during the testing session. An error is defined as a participant meeting one of the following criteria: moving the hands from the iPad, opening the eyes, step stumble or fall, abduction or flexion of the hip beyond 30°, lifting the forefoot or heel off of the testing surface, remaining out of the proper testing position for greater than 5 seconds. Each trial, or condition can have a maximum of 10 errors. If a subject commits multiple errors simultaneously, only one error is recorded. For example, if an individual steps or stumbles, opens their eyes, and removes their hands from their hips simultaneously, then they are credited with only one error.

ELIGIBILITY:
Inclusion Criteria:

* Must participate in at least 120 minutes of self-reported leisure-time physical activity.

Exclusion Criteria:

* Individual has had a concussion within the past 3 months
* Individual is currently going through rehabilitation for a musculoskeletal injury
* Individual has a known neurological disorder that would affect their balance (e.g. vertigo, meniere's disease)
* A female volunteer reports they are pregnant

Ages: 19 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Volunteers will be recruited from the University of Nebraska at Omaha campus community, and we aim to include both undergraduate and graduate students. The sample aims to reflect a young, uninjured, and physically active population.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Bland-Altman Analysis | through study completion, approximately 6 months
  Limits of agreement between measures and bias estimates will be calculated to determine the agreement between the 3 different balance measurement techniques.

SECONDARY OUTCOMES:
Sway Balance Score | Immediate
  Score between 0 and 100 from a proprietary algorithm. A score of 0 indicates poor balance based off of measured sway. A score of 100 indicates excellent balance based off of the measurement of postural sway from a smart phone.
Balance Error Scoring System | Immediate
  The Balance Error Scoring System is a subjective rating of errors during standing balance. Errors are marked when: moving the hands from the iPad, opening the eyes, step stumble or fall, abduction or hip flexion beyond 30°, lifting the forefoot or heel off the ground, being out of testing position for greater than 5 seconds.
Sample Entropy of the center of pressure | Immediate
  Non-linear measure of the tendency of a pattern of a given data length will repeat. Values range between 0 and 2. Values closer to 0 indicate highly regular and predictable signals with patterns. Values closer to 2 indicate less regular signals, with less predictability and more randomness. Analysis performed in MATLAB from the center of pressure data recorded from the Balance Tracking Systems force platform.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Burcal, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska at Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No